CLINICAL TRIAL: NCT02682043
Title: Parental Perspectives of Using Modified Toy Cars on the Social Interactions of Preschool Children With Mobility Impairments.
Brief Title: Parental Perspectives of Using Toy Cars on Social Interactions of Preschool Children With Mobility Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 15/0131
Record Dates: First submitted 2016-01-26; First posted 2016-02-15 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-09

CONDITIONS: Children; Mobility Limitation; Spina Bifida; Attitude to Health
MeSH Terms: conditions — Mobility Limitation; Spinal Dysraphism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Toy car (Experimental): The intervention is the provision of an electric toy car. This toy car will be modified to meet the postural and hand control preference of each child participant.
  Interventions: Device: Toy car

INTERVENTIONS:
Device: Toy car — The intervention is the provision of an electric toy car. This toy car will be modified to meet the postural and hand control preference of each child participant.
  The child will have the toy car for an 8 week trial period. Parents and child will be instructed in the safe use of the toy car, given written guidelines, and encouraged to use frequently.
  Parents will keep a log of what days they use the toy car, where and for how long.

SUMMARY:
The purpose of this study is to investigate parental attitudes towards their child who has a mobility impairment, to using a modified electric toy car, and to evaluate from their perspective, if it facilitated social interaction for their child with mobility impairment.

DETAILED DESCRIPTION:
Project Aims:

The overall aim of the project is to investigate parental perspectives on the impact of using a modified electric toy car on social interactions of pre-school children with mobility impairments, over an 8 week period.

A secondary aim is to understand from the parent's perspective, features of the toy car they valued and features they feel could be changed to improve the experience for their child.

Methods:

Participants will be recruited via a charity in Northern Ireland who supports parents of children with Spina Bifida who have mobility impairments (SHINE). Once participants are confirmed, they will attend clinic appointments at Musgrave Park Hospital, Belfast. At clinic, the principle investigator will complete an assessment of the child to determine what modifications are required to support the child in the toy car as well as modifications to access drive functions.

The participants will be shown 3 possible toy car options and the child will have the opportunity to try driving the cars. Parents will then select the toy car they wish to use allowing them to consider aesthetic features. Giving the parents the option of selecting the car enhances patient and public involvement in the study.

Following this, the car will be ordered and modifications completed. The rehabilitation engineer will complete a medical device risk assessment on each car to ensure safety. A second appointment will then evaluate modifications, complete final adjustments and a safety handover.

Parents will be asked to use the toy car during social interactions with the child over an 8 week period. They will be asked to keep a log of their experiences over this time. Following this, the principle investigator will complete semi-structured interviews with the parents to determine their experiences of using the toy car.

Sample size: 5 child participants aged between 12 months and 47 months.

Outcome measures: Semi structured interviews will be completed with parents after 8 week trial intervention. In addition the PIADS will be completed before and after the trial to see if this can predict the likelihood for the parents to use the modified toy car, and what impact it has on their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 12 months and 3 years, 11 months.
* Parents or Guardians aged 18 years and over, fluent English language speakers.
* Children who are unable to walk independently.
* Children who have no experience of using powered wheelchairs.
* Children who do not have a diagnosed severe learning disability.
* Children, who are medically stable, do not require ventilation or suction and can maintain upright head positioning when seated on a flat surface.

Exclusion Criteria:

* Children with a diagnosis of severe learning disability.
* Children, who are currently medically unwell, require ventilation, suction and can't maintain an upright head position when seated on a flat surface.

Ages: 12 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Parent Interview | on completion of 8 week trial
  Semi-structured interview investigating impact on child's play and social experiences, reactions of child and others; barriers to using car; parent response and emotions to child using car; ideas to improve the experience; would they/child continue to use the toy car.

SECONDARY OUTCOMES:
Psychosocial Impact of Assistive Devices Scale (PIADS) - Jutai & Day 2002 | Baseline and on completion of 8 week trial
  Standardised Questionnaire used to determine if the assistive device improves the perceived quality of life of users; and can predict the retention or abandonment of the device.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Casey, MSc, Study Chair — University of Ulster; Laura McKeown, PhD, Study Chair — University of Ulster

IPD SHARING:
Plan to Share IPD: Yes
On completion of study - data will be analyzed and disseminated through paper/ conference presentations. All data will be anonymized.